CLINICAL TRIAL: NCT01062997
Title: Volar Locked Plating Versus Bridging External Fixation
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Ola-Lars Hammer, PhD-student, University Hospital, Akershus
Other Study IDs: S-09101a 2009/2172
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
A randomized, prospective comparison of volar locked plating versus Hoffman II bridging external fixation supplemented by K-wire fixation in patients with comminuted distal radius fractures, AO/OTA type C2 & C3.

Hypothesis:

There is no significant difference in using volar plates compared to Hoffman II bridging external fixation supplemented by K-wire fixation in patients with comminuted distal radius fractures, AO/OTA type C2 & C3 as evaluated by a Quick-DASH score at 24 months follow-up.

DETAILED DESCRIPTION:
We have designed a randomized, prospective study for comparison of volar locked plating versus Hoffman II bridging external fixation supplemented by K-wire fixation in patients with comminuted distal radius fractures, AO/OTA type C2 & C3. On the basis of power analysis a total of 140 patients are to be included in this project. The follow-up period is 2 years and evaluation is based on x-ray analysis, grip strength, range of movement, pain and various tools to measure quality of life and satisfaction with the treatment (EQ-5d, SF-36, Quick-DASH).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Ahus and Lillestrom legevakt with a distal radius fracture are to be classified according to the system of the Orthopaedic Trauma Association (AO/OTA).
* All patients between the age of 18 and 70 diagnosed with a C2- or C3-type fracture, or a dislocated C1-fracture, are eligible for inclusion.

Exclusion Criteria:

* Gustillo-Anderson type III open fractures
* Previous distal radius/ulna-fracture and/or disabling hand injury of the same extremity
* Dementia
* Congenital anomaly
* Bilateral radius fracture
* Pathological fracture other than osteoporotic fracture
* Congenital bone disease (for example osteogenesis imperfecta)
* Age below 18 and above 70
* Disabling nury to other parts og the movement apparatus at the same time as the current injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between the age of 18 and 70 diagnosed with a C2- or C3-type fracture
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quick-DASH | 2 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Sykehusveien 25, Nordbyhagen, Lorenskog, Norway